CLINICAL TRIAL: NCT01329744
Title: Effects of Recombinant IGF-I in HIV Associated Metabolic Disease
Brief Title: Effects of IGF-I in HIV Metabolic Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Roy Kim, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1K23DK080644-01A1 (NIH)
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: HIV Lipodystrophy
Keywords: HIV lipodystrophy
MeSH Terms: interventions — mecasermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Recombinant IGF-I
  Interventions: Drug: mecasermin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: mecasermin — a subcutaneous injection twice a day
  Other Names: Increlex
  Arms: Treatment
Drug: Placebo control — Subcutaneous injection given twice per day of placebo compound, for 24 weeks
  Arms: Placebo

SUMMARY:
This study examines the effects of recombinant insulin like growth factor - I on body composition, glucose homeostasis, and lipids, in adults with HIV infection and signs of metabolic disease.

DETAILED DESCRIPTION:
The main objectives of this study are the following:

1. Determine the effect of recombinant human insulin like growth factor-I (rhIGF-I) (generic: mecasermin) on subcutaneous adiposity in patients with HIV lipodystrophy syndrome.
2. Determine the effects of rhIGF-I on glucose homeostasis and lipids in patients with HIV lipodystrophy.
3. Determine the effects of rhIGF-I on apoptosis, mitochondria, and inflammation, in adipose tissue obtained from patients with HIV lipodystrophy.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive with undetectable viral load
* No change in antiretrovirals for 3 months
* Evidence of lipoatrophy in the limbs, and face or gluteal area
* Dyslipidemia defined as:
* Fasting triglycerides > 200 OR
* HDL cholesterol < 40 mg/dL
* Abnormal glucose homeostasis defined as:
* Fasting hyperinsulinemia > 20 uU/mL OR
* Fasting glucose 100-125 mg/dL, inclusive

Exclusion Criteria:

* Two consecutive viral >75 or > 50 copies/mL using the tests listed above
* Presence of AIDS wasting
* Change in antiretroviral medication (not dose) in the prior 3 months
* Coronary artery disease, cerebrovascular, or peripheral arterial disease
* Diabetes mellitus
* Adrenal insufficiency, hypoglycemia, thyroid disease, or other endocrine disorder that is untreated
* Malignancy
* Eating disorder
* Pregnancy (urine pregnancy test is required of all females)
* Previous liposuction or bariatric surgery
* Other systemic conditions or other disorders at the discretion of the investigators
* Current use of systemic glucocorticoids, or other agent affecting body weight or glucose homeostasis or other drug at the discretion of the investigators
* Use of interferon within the past six months
* Use of insulin, insulin secretagogue, thiazolidinedione, or metformin in the prior 3 months
* Initiation or dose adjustment, within the prior 3 months, of any of the following drugs or drug classes: fibrate, cholesterol binding resin, statin, niacin, or omega 3 fatty acid (fish oil).
* Use of uridine, growth hormone, IGF-I, and growth hormone releasing factor analogues

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Body composition | 24 weeks
  Participants will have a body scan called a dual energy x-ray absorptiometry (DEXA) scan and a single slice abdominal CT scan and mid thigh scan to measure subcutaneous and internal fat.

SECONDARY OUTCOMES:
Glucose Homeostasis | 24 weeks
  Fasting glucose and insulin will be measured. A subset of patients will undergo a hyperinsulinemic clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Roy J Kim, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States